CLINICAL TRIAL: NCT04862949
Title: Organ-specific Responses to Atezolizumab Plus Bevacizumab in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Organ-specific Responses to Atezolizumab Plus Bevacizumab in Advanced HCC
Status: Completed | Type: Observational
Sponsor: CHA University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-04-010-001
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma, atezolizumab, bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atezolizumab plus bevacizumab: Patients received combination therapy with atezolizumab and bevacizumab as first-line systemic treatment for advanced HCC.
  Interventions: Drug: Atezolizumab plus bevacizumab

INTERVENTIONS:
Drug: Atezolizumab plus bevacizumab — Patients received combination therapy with atezolizumab (Tecentriq) and bevacizumab (Avastin) as first-line systemic treatment for advanced hepatocellular carcinoma.
  Other Names: Atezolizumab; Bevacizumab

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most frequent causes of cancer-related deaths globally and in Korea. Many patients diagnosed at advanced stage, and systemic therapy is mainstay of treatment in patients with advanced HCC.

However, immune-checkpoint inhibitor (ICI) monotherapy did not significantly improve overall survival in phase III studies. According to previous retrospective analyses, ICI treatment in advanced HCC showed different organ-specific responses. The intrahepatic HCC was the least responsive organ to ICI treatment. The failure of phase III trials of ICI monotherapy may have been attributed to different organ-specific response pattern of ICIs.

Combination of atezolizumab plus bevacizumab is expected to overcome the immunosuppressive microenvironment of liver and may enhance intrahepatic response of ICI.

DETAILED DESCRIPTION:
In a previous retrospective analysis of pembrolizumab treated patients with advanced melanoma and NSCLC, patients with liver metastases showed poorer PFS compared with those without liver metastases with reduced ORR. Similar observations have also been reported in metastatic of triple-negative breast cancer patients, there were no responses in patients with liver metastases. Taken together the results of previous studies, hepatic metastases had reduced response to ICI compared with metastases at other organs, regardless of cancer types.

In addition, ICI treatment in advanced HCC showed different organ-specific responses. The poorer response rate in liver to ICI might be affected by liver-specific immunosuppressive microenvironment (TME). To overcome the unfavorable immunosuppressive TME of the liver, combination strategies are needed to achieve enhanced anti-tumor immune responses or alleviated tumor-associated immunosuppression.

Since the cause of death in most HCC patients was hepatic failure due to intrahepatic HCC or underlying liver cirrhosis, the response rate to ICI of intrahepatic tumor lesions is a crucial factor in determining the overall prognosis of advanced HCC.

Therefore, we hypothesize that combination strategy of atezolizumab plus bevacizumab may increase organ specific response in patients with advanced HCC, and may improve survival outcomes accordingly.

Objectives We hypothesize that combination strategy of atezolizumab plus bevacizumab may increase organ specific response in patients with advanced HCC, and may improve survival outcomes accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HCC pathological or non-invasive assessment according to American Association for the Study of Liver Diseases (AASLD) criteria
* ECOG performance status 0 or 1
* Patients who received Atezolizumab and Bevacizumab combination therapy as first-line systemic treatment for unresectable HCC
* Barcelona Clinic Liver Cancer (BCLC) stage B or C
* Child-Pugh class A
* Measurable lesion
* Adequate hematologic and organ function

Exclusion Criteria:

* History of autoimmune disease
* Concomitant anticoagulation at therapeutic doses. Low dose aspirin for
* cardio protection is permitted.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrollment was performed in the CHA Bundang Medical Center, Ulsan University Hospital and Chinese University of Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD, PhD, Principal Investigator — CHA University
Locations (1):
- Cha Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Montal R, Sia D, Finn RS. Molecular therapies and precision medicine for hepatocellular carcinoma. Nat Rev Clin Oncol. 2018 Oct;15(10):599-616. doi: 10.1038/s41571-018-0073-4. PMID 30061739
- [Background] Jung KW, Won YJ, Oh CM, Kong HJ, Lee DH, Lee KH; Community of Population-Based Regional Cancer Registries. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2014. Cancer Res Treat. 2017 Apr;49(2):292-305. doi: 10.4143/crt.2017.118. Epub 2017 Mar 9. PMID 28279062
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Background] Lu LC, Hsu C, Shao YY, Chao Y, Yen CJ, Shih IL, Hung YP, Chang CJ, Shen YC, Guo JC, Liu TH, Hsu CH, Cheng AL. Differential Organ-Specific Tumor Response to Immune Checkpoint Inhibitors in Hepatocellular Carcinoma. Liver Cancer. 2019 Nov;8(6):480-490. doi: 10.1159/000501275. Epub 2019 Aug 6. PMID 31799205
- [Background] Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, Latreche S, Bergaya S, Benhamouda N, Tanchot C, Stockmann C, Combe P, Berger A, Zinzindohoue F, Yagita H, Tartour E, Taieb J, Terme M. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med. 2015 Feb 9;212(2):139-48. doi: 10.1084/jem.20140559. Epub 2015 Jan 19. PMID 25601652
- [Background] Motz GT, Santoro SP, Wang LP, Garrabrant T, Lastra RR, Hagemann IS, Lal P, Feldman MD, Benencia F, Coukos G. Tumor endothelium FasL establishes a selective immune barrier promoting tolerance in tumors. Nat Med. 2014 Jun;20(6):607-15. doi: 10.1038/nm.3541. Epub 2014 May 4. PMID 24793239
- [Background] Hegde PS, Wallin JJ, Mancao C. Predictive markers of anti-VEGF and emerging role of angiogenesis inhibitors as immunotherapeutics. Semin Cancer Biol. 2018 Oct;52(Pt 2):117-124. doi: 10.1016/j.semcancer.2017.12.002. Epub 2017 Dec 8. PMID 29229461
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Pao W, Ooi CH, Birzele F, Ruefli-Brasse A, Cannarile MA, Reis B, Scharf SH, Schubert DA, Hatje K, Pelletier N, Spleiss O, Reed JC. Tissue-Specific Immunoregulation: A Call for Better Understanding of the "Immunostat" in the Context of Cancer. Cancer Discov. 2018 Apr;8(4):395-402. doi: 10.1158/2159-8290.CD-17-1320. Epub 2018 Mar 15. PMID 29545369
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Tumeh PC, Hellmann MD, Hamid O, Tsai KK, Loo KL, Gubens MA, Rosenblum M, Harview CL, Taube JM, Handley N, Khurana N, Nosrati A, Krummel MF, Tucker A, Sosa EV, Sanchez PJ, Banayan N, Osorio JC, Nguyen-Kim DL, Chang J, Shintaku IP, Boasberg PD, Taylor EJ, Munster PN, Algazi AP, Chmielowski B, Dummer R, Grogan TR, Elashoff D, Hwang J, Goldinger SM, Garon EB, Pierce RH, Daud A. Liver Metastasis and Treatment Outcome with Anti-PD-1 Monoclonal Antibody in Patients with Melanoma and NSCLC. Cancer Immunol Res. 2017 May;5(5):417-424. doi: 10.1158/2326-6066.CIR-16-0325. Epub 2017 Apr 14. PMID 28411193
- [Background] Adams S, Schmid P, Rugo HS, Winer EP, Loirat D, Awada A, Cescon DW, Iwata H, Campone M, Nanda R, Hui R, Curigliano G, Toppmeyer D, O'Shaughnessy J, Loi S, Paluch-Shimon S, Tan AR, Card D, Zhao J, Karantza V, Cortes J. Pembrolizumab monotherapy for previously treated metastatic triple-negative breast cancer: cohort A of the phase II KEYNOTE-086 study. Ann Oncol. 2019 Mar 1;30(3):397-404. doi: 10.1093/annonc/mdy517. PMID 30475950
- [Background] Gao Q, Qiu SJ, Fan J, Zhou J, Wang XY, Xiao YS, Xu Y, Li YW, Tang ZY. Intratumoral balance of regulatory and cytotoxic T cells is associated with prognosis of hepatocellular carcinoma after resection. J Clin Oncol. 2007 Jun 20;25(18):2586-93. doi: 10.1200/JCO.2006.09.4565. PMID 17577038
- [Background] Eggert T, Greten TF. Tumor regulation of the tissue environment in the liver. Pharmacol Ther. 2017 May;173:47-57. doi: 10.1016/j.pharmthera.2017.02.005. Epub 2017 Feb 4. PMID 28167218
- [Background] Hoechst B, Ormandy LA, Ballmaier M, Lehner F, Kruger C, Manns MP, Greten TF, Korangy F. A new population of myeloid-derived suppressor cells in hepatocellular carcinoma patients induces CD4(+)CD25(+)Foxp3(+) T cells. Gastroenterology. 2008 Jul;135(1):234-43. doi: 10.1053/j.gastro.2008.03.020. Epub 2008 Mar 21. PMID 18485901
- [Background] Ji J, Eggert T, Budhu A, Forgues M, Takai A, Dang H, Ye Q, Lee JS, Kim JH, Greten TF, Wang XW. Hepatic stellate cell and monocyte interaction contributes to poor prognosis in hepatocellular carcinoma. Hepatology. 2015 Aug;62(2):481-95. doi: 10.1002/hep.27822. Epub 2015 Apr 28. PMID 25833323
- [Background] Berg M, Wingender G, Djandji D, Hegenbarth S, Momburg F, Hammerling G, Limmer A, Knolle P. Cross-presentation of antigens from apoptotic tumor cells by liver sinusoidal endothelial cells leads to tumor-specific CD8+ T cell tolerance. Eur J Immunol. 2006 Nov;36(11):2960-70. doi: 10.1002/eji.200636033. PMID 17039564
- [Background] Wu Y, Kuang DM, Pan WD, Wan YL, Lao XM, Wang D, Li XF, Zheng L. Monocyte/macrophage-elicited natural killer cell dysfunction in hepatocellular carcinoma is mediated by CD48/2B4 interactions. Hepatology. 2013 Mar;57(3):1107-16. doi: 10.1002/hep.26192. Epub 2013 Jan 18. PMID 23225218
- [Background] Li H, Wu K, Tao K, Chen L, Zheng Q, Lu X, Liu J, Shi L, Liu C, Wang G, Zou W. Tim-3/galectin-9 signaling pathway mediates T-cell dysfunction and predicts poor prognosis in patients with hepatitis B virus-associated hepatocellular carcinoma. Hepatology. 2012 Oct;56(4):1342-51. doi: 10.1002/hep.25777. PMID 22505239
- [Background] Uka K, Aikata H, Takaki S, Shirakawa H, Jeong SC, Yamashina K, Hiramatsu A, Kodama H, Takahashi S, Chayama K. Clinical features and prognosis of patients with extrahepatic metastases from hepatocellular carcinoma. World J Gastroenterol. 2007 Jan 21;13(3):414-20. doi: 10.3748/wjg.v13.i3.414. PMID 17230611
- [Background] Cheon J, Jung S, Kim JS, Kang B, Kim H, Chan LL, Becker L, Gaillard VE, Chan SL, Kim C, Chon HJ. Organ-specific responses to atezolizumab plus bevacizumab in advanced hepatocellular carcinoma: A multicentre, retrospective study. Liver Int. 2024 Aug;44(8):1961-1970. doi: 10.1111/liv.15935. Epub 2024 Apr 15. PMID 38618972
- See also: Lee M, Ryoo BY, Hsu CH, et al: Randomised efficacy and safety results for atezolizumab (Atezo) + bevacizumab (Bev) in patients (pts) with previously untreated, unresectable hepatocellular carcinoma (HCC). Annals of Oncology 30:v875, 2019 — https://pubmed.ncbi.nlm.nih.gov/31559039/
- See also: T. Yau, J.W. Park, R.S. Finn, et al: LBA38_PR - CheckMate 459: A randomized, multi-center phase III study of nivolumab (NIVO) vs sorafenib (SOR) as first-line (1L) treatment in patients (pts) with advanced hepatocellular carcinoma (aHCC). — https://doi.org/10.1093/annonc/mdz394.029

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab Plus Bevacizumab: Atezolizumab plus bevacizumab
  Atezolizumab plus bevacizumab: Atezolizumab plus bevacizumab
Period: Overall Study
Arm/Group | Atezolizumab Plus Bevacizumab
Started | 131
Completed | 131
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We enrolled patients who received first-line Ate/Bev treatment for aHCC. Eligible patients included those with Child-Pugh A liver function, measurable tumor lesions, and serial image studies available for response evaluation.
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 131
Age, Continuous [Median (Full Range); unit: years]
  Age | 62 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 110
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race and Ethnicity data were not collected in this study (South Korea, Hong Kong).
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 131
Region of Enrollment [Number; unit: participants]
  South Korea | 124
  Hong Kong | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lesions With Organ-specific Response
Description: Organ-specific response will be assessed at the lesion level according to RECIST 1.1 criteria. Up to two target lesions per organ (maximum of five total lesions per patient) will be selected and measured unidimensionally. Complete response (CR) is defined as disappearance of the lesion or lymph node short axis diameter <1.0 cm. Partial response (PR) is defined as ≥30% reduction in lesion size. Progressive disease (PD) is defined as ≥20% increase in lesion size. Stable disease (SD) is defined as neither CR, PR, nor PD. New lesions are recorded in addition to original target lesions to determine the total tumor burden.
Time Frame: From treatment initiation until last follow-up (median 10.1 months)
Population: Organ-specific responses were assessed for 260 individual tumor lesions from 131 participants who received atezolizumab plus bevacizumab: 152 liver lesions, 42 lymph node lesions, 24 lung lesions, and 42 other metastatic lesions were evaluated.
Measure: Number; unit: Percentage of Units (lesions)
Units Other Than Participants: lesion
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 131
Number analyzed (lesion) | 260
Percentage of Units (lesions)
  ORR for 260 individual tumor lesions | 29.8
  ORR for 152 liver lesions: number analyzed (lesion) | 152
  ORR for 152 liver lesions | 28.3
  ORR for 42 LNs lesions: number analyzed (lesion) | 42
  ORR for 42 LNs lesions | 40.5
  ORR for 24 lungs lesions: number analyzed (lesion) | 24
  ORR for 24 lungs lesions | 29.1
  ORR for other metastatic lesions: number analyzed (lesion) | 42
  ORR for other metastatic lesions | 19.0

ADVERSE EVENTS:
Time Frame: From treatment initiation until last follow-up (median 10.1 months)
Description: Adverse events were collected from the start of treatment until last follow-up, and were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
Arm/Group | Atezolizumab Plus Bevacizumab
All-Cause Mortality (participants affected / at risk) | 57/131
Serious Adverse Events (participants affected / at risk) | 16/131
Other Adverse Events (participants affected / at risk) | 108/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Plus Bevacizumab (N=131)
Gastrointestinal bleeding (Grade ≥3) (Gastrointestinal disorders) | 6 (6)
Proteinuria (Grade ≥3) (Renal and urinary disorders) | 3 (3)
Hypertension (Grade ≥3) (Vascular disorders) | 3 (3)
Other treatment-related SAEs (General disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Plus Bevacizumab (N=131)
Fatigue (General disorders) | 26 (26)
Decreased appetite (Metabolism and nutrition disorders) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12)
Proteinuria (Renal and urinary disorders) | 15 (15)
Hypertension (Vascular disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT04862949/Prot_SAP_000.pdf